CLINICAL TRIAL: NCT05758792
Title: Does Poor Muscle Quality in Older Women Affect Fall Concern and Lower Extremity Functionality?
Brief Title: Muscle Quality, Fall Concern and Lower Extremity Functionality in Older Women
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Güzin Kara, PT., PhD., Pamukkale University
Other Study IDs: 60116787-020/71654
Record Dates: First submitted 2022-11-25; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Old Age; Debility; Age-Related Sarcopenia
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Muscle Quality Index — Evaluations are applied to older adults to compare the results of muscle quality.
  Other Names: Lower Extremity Functional Scale; International Fall Efficiency Scale

SUMMARY:
The aim of the study was to investigate the effects of muscle quality on fear of fall, and lower extremity functionality in older women. The differences between muscle quality, fear of falling and lower extremity functionality in the elderly male and female participating in the study were investigated. Older women had worse muscle quality, higher fall concern and less lower extremity functionality than older men.

DETAILED DESCRIPTION:
The effects of muscle quality and lower extremity functionality, and fear of falling in older women are not well-known compared to older men in the same age group. The aim of the study was to investigate the effects of muscle quality on lower extremity functionality and fear of falling in older women. 168 age-matched older adults participated in the study. The muscle quality Index, fear of fall, and lower extremity functionality were evaluated. The results of older women and men were compared.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years old or older
* Having no neurological, orthopedic, communicational,
* Mental disability that affects the evaluations.

Exclusion Criteria:

* Incomplete data and older adults not agreeing to participate in the study.

Ages: 65 Years to 85 Years | Sex: All
Age Groups: Older Adult
Gender Based: Yes — This study was planned to investigate the effects of muscle quality on older women comparing to older men.
Study Population: Age-matched older men and women were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Muscle Quality Index | 6 months
  Muscle Quality Index scored is calculated through anthropometric measurements of older adults. The muscle quality depends on the formula as follows: MQI (Watts) = ((Leg length×0.4)×Body mass×gravity ×10)/ Five Times Sit To Stand.
Lower Extremity Functional Scale | 6 months
  LEFS presents 20 questions about daily living activities. The questionnaire was developed to assess lower extremity functionality and can be used in older adults.The minimum and maximum total score ranges from 0 to 80. High scores show high functional status.
International Fall Efficiency Scale | 6 months
  The scale consist of items about fall concern during daily living activities. The minimum and maximum total score ranges from 16 to 64. High scores represents high fall concern.

CONTACTS AND LOCATIONS:
Overall Officials: Güzin Kara Çakıcı, PhD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data.

REFERENCES:
- [Result] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Result] Fragala MS, Fukuda DH, Stout JR, Townsend JR, Emerson NS, Boone CH, Beyer KS, Oliveira LP, Hoffman JR. Muscle quality index improves with resistance exercise training in older adults. Exp Gerontol. 2014 May;53:1-6. doi: 10.1016/j.exger.2014.01.027. Epub 2014 Feb 6. PMID 24508922
- [Result] Gadelha AB, Neri SGR, Nobrega OT, Pereira JC, Bottaro M, Fonseca A, Lima RM. Muscle quality is associated with dynamic balance, fear of falling, and falls in older women. Exp Gerontol. 2018 Apr;104:1-6. doi: 10.1016/j.exger.2018.01.003. Epub 2018 Jan 9. No abstract available. PMID 29329971